CLINICAL TRIAL: NCT03559712
Title: Effectiveness of Collaborative Tele-Mental Health Services for ADHD in Primary Care: A Randomized Trial in Dubai (ECTSAP- Dubai Trial)
Brief Title: Effectiveness of Collaborative Tele-Mental Health Services for ADHD in Primary Care
Acronym: ECTSAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Jalila Children's Specialty Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Dr. Ammar AlBanna, Head of Child and Adolescent Mental Health Center of Excellence, Consultant Child and Adolescent Psychiatrist, Al Jalila Children's Specialty Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 027562-746845-0105
Record Dates: First submitted 2018-05-24; First posted 2018-06-18 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: ADHD; Telemental Health
Keywords: Attention Deficit Hyperactivity Disorder; Collaborative Care; Telemedecine; Telemental Health
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Using a collaborative care approach with the aid of telemedicine to treat children with ADHD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Participants in this arm will be treated by the trained primary health care physicians in the primary health care centers, who will be having weekly supervisions with the specialists for case management.
  Interventions: Other: Collaborative care, Telemental health
- Control (No Intervention): Participants in this arm will experience treatment as usual, which means referral to a specialist.

INTERVENTIONS:
Other: Collaborative care, Telemental health — Children who are referred to the collaborative tele-mental health care arm, Arm (1), will be given a follow-up appointment with the physician at the same primary care center who have successfully completed the pre-trial didactic program designed by Drs. Albanna and Hamoda. The trained child health physician will conduct assessments, treat and manage the patient. All while having weekly clinical supervision with the specialist.
  Arms: Telemedicine

SUMMARY:
Aim and objectives:

In this study, our goal is to assess the effectiveness of a collaborative tele-mental health approach for treatment of children and adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD) presenting to primary healthcare centers in Dubai.

Our primary aim is:

To determine if collaborative tele-mental health program improves the clinical and functional outcomes for children with Attention-deficit/hyperactivity disorder (ADHD) in Dubai

Secondary aims:

1. To improve the ability of primary health-care providers to diagnose and treat pediatric ADHD, leading to enhanced community capacity, improving patient access and ensuring sustainability.
2. To enhance parent and child satisfaction with the ADHD assessment and treatment process in Dubai.

DETAILED DESCRIPTION:
Potential Significance:

There are presently very limited clinical resources for children with ADHD, a prevalent disorder associated with significant functional impairments across different domains. Given the large number of affected children and their families, and the lack of readily available resources, very long wait-lists exist delaying access to healthcare. This is especially important given that ADHD occurs during a critical period of child development. Despite that effective treatments for ADHD do exist, it is quite challenging to deliver timely interventions to children with ADHD. This study aims to assess the efficacy of an innovative collaborative care approach that significantly improves access to evidence based health services and builds capacity in the community. Given that public healthcare services in Dubai are open to all emirates in the UAE and that some specialized services are lacking in other emirates, such a program that utilizes a virtual platform will facilitate healthcare access to this group of children in remote areas. After providing evidence for its feasibility and efficacy, this approach is likely to then be implemented across Dubai's Health Authority and to become a model that can be implemented nationally and regionally.

This study will significantly enhance the capacity of primary care physicians in Dubai, UAE to provide clinical care for children with common mental health conditions, namely ADHD. Enhancing the capacity of the Primary care sector to assess and treat this disorder in collaboration with the center of excellence at Al Jalila Children's is expected to improve access to clinical care while assuring optimal care is provided.

Moreover, it will improve the expertise of the center of excellence in child mental health at Al Jalila children's through clinical and research collaboration with Boston Children's Hospital. This study might open the doors for future collaborations with international institute such Boston Children's which will result in improved pediatric care at Al Jalila Children's. After providing evidence for its feasibility and efficacy, this approach is likely to then be implemented across Dubai's Health Authority and to become a model that can be implemented nationally and regionally.

Methods:

An individually randomized controlled trial with 2 equal groups will be conducted. Children aged 6-12 years who are referred to their primary care provider for an ADHD assessment and meet inclusion criteria will be randomized to intervention and control arms.

The intervention will consist of treatment of children with ADHD by physicians trained by study staff on the assessment and treatment of ADHD. This training will be delivered over two stages:

In stage (1), prior to any clinical interaction with patients, physicians will attend an on-site clinical training that includes didactic teaching on ADHD including reviewing clinical guidelines and hands-on assessment and treatment of children with ADHD presenting to the tertiary care hospital (minimum of 35 hours). Drs. Albanna and Hamoda will deliver this training. Participants will be expected to successfully complete two PDM exam stations (Phenomenology, Diagnosis and Management). These PDM stations will be developed by AA and HH and will not include real patients. This educational intervention will be delivered prior to any interaction between pediatricians and patients, and only those pediatricians that successfully complete the course will participate in the collaborative-care arm of the study.

In stage (2) of the training program, an ongoing module will be developed by Drs. Albanna and Hamoda using a virtual-classroom setup. This will include monthly live online presentations presented by Drs. Albanna and Hamoda as well as invited guest speakers for select topic, that Drs. Albanna and Hamoda will moderate. This intends to discuss advanced topics and challenges that may be facing the clinicians involved in the study. The research coordinator will assure that the technical setup is prepared for the seminars. There will be a total of 8 presentations, and the duration will be 1 and half hours for each presentation. The topics will focus on various advanced aspects of managing ADHD in primary healthcare. Pre-presentation reading material will be emailed to the attendees along with details regarding the time and topic of the presentation. They will be asked to log-on 15 minutes prior and the last 30 minutes will be dedicated to discussions and questions relevant to the topic. Every presentation will be followed by 10 MCQs prepared by the presenter. Participants will also have weekly supervision meetings via video-conferencing. Randomization will occur when children with suspected ADHD present to PHCs participating in this study. Children will be randomly referred to one of these two study arms:

Arm (1): Children in this arm will received a collaborative mental health model of care by physicians who underwent the training above. Children and their families will be assessed and managed by these physicians, at the same primary care center they present at, using international guidelines. In line with the collaborative care model, physicians in this arm will have weekly supervision meetings via video-conferencing with specialists from the study team. Case management will be provided via trained allied professional or nurse. Case management will entail assuring that patients present on time for scheduled assessment and follow-ups and that questionnaires are completed and handed on time.

Arm (2): The children randomized to control arm will receive treatment as usual. This primarily consists of referral to specialized mental health services at Al Jalila Children's. They will receive assessment and management by specialists in this tertiary care center.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6-12 years
* Children who meet DSM-5 criteria for ADHD as determined by both clinical assessment and the Vanderbilt ADHD scales.

Exclusion Criteria:

* Active clinically significant medical illness (e.g. cardiac and seizure disorders).
* Family history of early onset cardiac disease.
* Autism spectrum disorder or clinically significant developmental delay.
* Intellectual disability (IQ of 70 and below, or diagnosis of intellectual disability).
* Active primary psychiatric illness other than ADHD (e.g. mood disorder, anxiety disorder, psychotic disorder, tic disorder).
* Previous ADHD diagnosis and treatment.
* Currently taking psychiatric medications for any indication.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
NIHCQ Vanderbilt assessment scale (Parent) | At baseline, 3-month follow-up and 6-month follow-up
  Change in Total Symptom Score for ADHD symptoms in Vanderbilt parent informant form and follow-up forms (at 3 and 6-months follow-up)

CONTACTS AND LOCATIONS:
Locations (2):
- United Arab Emirates (2):
  - Dubai Health Authority, Dubai
  - Al Jalila Children's Specialty Hospital, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eapen V, Mabrouk AA, Zoubeidi T, et al. (2009) Epidemiological Study of Attention Deficit Hyperactivity Disorder Among School Children in the United Arab Emirates. HAMDAN MEDICAL JOURNAL, 2(3):119-127-127. doi:10.2174/1996327000902030119
- [Background] Myers K, Vander Stoep A, Lobdell C. Feasibility of conducting a randomized controlled trial of telemental health with children diagnosed with attention-deficit/hyperactivity disorder in underserved communities. J Child Adolesc Psychopharmacol. 2013 Aug;23(6):372-8. doi: 10.1089/cap.2013.0020. PMID 23952183
- [Background] Myers K, Vander Stoep A, Zhou C, McCarty CA, Katon W. Effectiveness of a telehealth service delivery model for treating attention-deficit/hyperactivity disorder: a community-based randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2015 Apr;54(4):263-74. doi: 10.1016/j.jaac.2015.01.009. Epub 2015 Jan 29. PMID 25791143
- [Background] Silverstein M, Hironaka LK, Walter HJ, Feinberg E, Sandler J, Pellicer M, Chen N, Cabral H. Collaborative care for children with ADHD symptoms: a randomized comparative effectiveness trial. Pediatrics. 2015 Apr;135(4):e858-67. doi: 10.1542/peds.2014-3221. PMID 25802346
- [Background] Epstein JN, Langberg JM, Lichtenstein PK, Altaye M, Brinkman WB, House K, Stark LJ. Attention-deficit/hyperactivity disorder outcomes for children treated in community-based pediatric settings. Arch Pediatr Adolesc Med. 2010 Feb;164(2):160-5. doi: 10.1001/archpediatrics.2009.263. PMID 20124145